CLINICAL TRIAL: NCT04106050
Title: A Phase 1b, Randomized, Double-Blind, Parallel, Placebo- and Active-Controlled, Pharmacodynamic Study of BIIB095 and BIIB074 in Healthy Participants and Participants With Painful Diabetic Polyneuropathy
Brief Title: Pharmacodynamic Study of BIIB095 and BIIB074 in Healthy Participants and Participants With Painful Diabetic Polyneuropathy
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 255NP101; 2019-001900-39 (EudraCT Number)
Record Dates: First submitted 2019-09-25; First posted 2019-09-26 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Healthy Volunteers; Diabetic Neuropathies
MeSH Terms: conditions — Diabetic Neuropathies | interventions — vixotrigine; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Part A: BIIB095 Dose 1 (Experimental): Healthy participants and participants with DPN will receive oral dose of BIIB095 Dose 1 capsules from Day 1 to Day 8.
  Interventions: Drug: BIIB095
- Part A: BIIB095 Dose 2 (Experimental): Healthy participants and participants with DPN will receive oral dose of BIIB095 Dose 2 capsules from Day 1 to Day 8.
  Interventions: Drug: BIIB095
- Part A: BIIB095 Dose 3 (Experimental): Healthy participants and participants with DPN will receive oral dose of BIIB095 Dose 3 capsules from Day 1 to Day 8.
  Interventions: Drug: BIIB095
- Part A: BIIB095 Placebo (Placebo Comparator): Healthy participants and participants with DPN will receive oral dose of placebo matching BIIB095 capsules from Day 1 to Day 8.
  Interventions: Drug: Placebo
- Part A: Lidocaine (Active Comparator): Healthy participants and participants with DPN will receive single injection of lidocaine for partial nerve conduction block and single injection of lidocaine for skin infiltration on Day 8.
  Interventions: Drug: Lidocaine
- Part B: BIIB074 Dose 1 (Experimental): Healthy participants and participants with DPN will receive oral dose of BIIB074 Dose 1 tablets from Day 1 to Day 8.
  Interventions: Drug: BIIB074
- Part B: BIIB074 Placebo (Placebo Comparator): Healthy participants and participants with DPN will receive oral dose of placebo matching BIIB074 tablets from Day 1 to Day 8.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIIB095 — Administered as specified in the treatment arm.
  Arms: Part A: BIIB095 Dose 1; Part A: BIIB095 Dose 2; Part A: BIIB095 Dose 3
Drug: BIIB074 — Administered as specified in the treatment arm.
  Arms: Part B: BIIB074 Dose 1
Drug: Placebo — Administered as specified in the treatment arm.
  Arms: Part A: BIIB095 Placebo; Part B: BIIB074 Placebo
Drug: Lidocaine — Administered as specified in the treatment arm.
  Arms: Part A: Lidocaine

SUMMARY:
Part A: Primary objective is to determine the effects of BIIB095 on nerve excitability in healthy participants. Secondary and exploratory objectives include determining the effects of BIIB095 on nerve excitability in diabetic polyneuropathy (DPN) and assessing the safety, tolerability and pharmacokinetics of BIIB095.

Part B (optional): Equivalent objectives are pursued for BIIB074.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy participants must be in good health, as determined based on medical history and screening evaluations
* Participants with DPN

  * Must have a documented diagnosis of type 2 diabetes mellitus (DM)
  * Must have stable glycemic control
  * Must have at least clinical evidence of painful DPN
  * Pain related to DPN must be present for at least 6 months prior to screening
  * Average daily pain intensity over 7 consecutive days recorded during screening must be ≥ 4 on an 11-point numerical rating scale ranging from 0 (no pain) to 10 (worst pain imaginable)

Key Exclusion Criteria:

* Any neurologic or painful condition that could confound the interpretation of study results
* History of any clinically significant cardiac, hematologic, hepatic, immunologic, urologic, pulmonary, dermatologic, psychiatric, renal, or other major disease. This includes any clinically significant endocrinologic or neurologic disease other than DM or DPN.
* Use of local anesthetics or capsaicin for topical or regional treatment within 3 months prior to Screening.
* Systemic use of sodium channel inhibitors

Note: Other protocol-specific inclusion/exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09-30 (Estimated); Primary Completion 2022-01-21 (Estimated); Study Completion 2022-01-21 (Estimated)

PRIMARY OUTCOMES:
Change in Nerve Excitability from Baseline (Day 1) to Last Treatment Visit (Day 8) as Determined by Compound Muscle Action Potential Threshold Tracking (CMAP-TT) in the Median Nerve of Healthy Participants | Baseline (Day 1), Day 8

SECONDARY OUTCOMES:
Change in Sensory Nerve Excitability from Baseline (Day 1) to Last Treatment Visit (Day 8) as Determined by Sensory Nerve Action Potential Threshold Tracking (SNAP-TT) in the Median Nerve of Healthy Participants | Baseline (Day 1), Day 8
Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) | AEs: Day 1 up to Day 22; SAEs: Screening up to Day 22
Area Under the Curve from Time Zero to Time of the Last Measurable Concentration (AUClast) | Pre-dose, 1 hour (h), 1.5h, 3h, 6h and 8h post-dose on Day 8
Area Under the Curve within a Dosing Interval (AUCtau) | Pre-dose, 1 hour (h), 1.5h, 3h, 6h and 8h post-dose on Day 8
Maximum Observed Concentration (Cmax) | Pre-dose, 1 hour (h), 1.5h, 3h, 6h and 8h post-dose on Day 8
Trough Concentration (Ctrough) | Pre-dose, 1 hour (h), 1.5h, 3h, 6h and 8h post-dose on Day 8
Time to Reach Maximum Observed Concentration (Tmax) | Pre-dose, 1 hour (h), 1.5h, 3h, 6h and 8h post-dose on Day 8

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on http://clinicalresearch.biogen.com/
URL: https://vivli.org/